CLINICAL TRIAL: NCT04101669
Title: A Randomized, Multi-Center, Pivotal Efficacy and Safety Study Evaluating the RESET® System for Glycemic Improvement in Patients With Inadequately Controlled Type 2 Diabetes and Obesity
Brief Title: RESET System Pivotal Trial (Rev F)
Acronym: STEP-1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Morphic Medical Inc. (Industry)
Collaborators: Biostatistical Consulting, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18-1
Record Dates: First submitted 2019-09-20; First posted 2019-09-24 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Diabetes type2; Obesity
Keywords: Type 2 Diabetes; Obesity
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2 | interventions — salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: A multi-center, double-blinded, randomized, sham-controlled trial to evaluate the safety and effectiveness of the RESET System. Patients will be randomized 3 (RESET):1 (Sham).
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The Investigators include interventional gastroenterologists (GI) and endocrinologists. The GI team: MD, PA and site coordinator, as well as radiology personnel will not be masked, while the endocrinologist team: the MDs, PAs, site coordinators and nutritionists, will be masked. The patient is also masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- RESET (Experimental): Patients in ARM 1, will receive an upper endoscopy and will be treated with the RESET Liner
  Interventions: Device: RESET Liner
- Sham (Sham Comparator): Patients in Arm 2 will receive an upper endoscopy, but will not be treated with the RESET Liner.
  Interventions: Other: Sham

INTERVENTIONS:
Device: RESET Liner — The RESET System is provided as a single-use, sterile device and consists of an RESET Liner preloaded, packaged and sterilized within the RESET Delivery System. The RESET Delivery System is utilized to deliver the RESET Liner to the proximal small intestine. The RESET Liner is removed using the RESET Retrieval System. The RESET System incorporates no pharmacological, biological tissue or blood products.
  Other Names: RESET Sleeve; Duodenal-jejunal Bypass Liner (DJBL); EndoBarrier
  Arms: RESET
Other: Sham — Patient receives upper endoscopy but no treatment
  Arms: Sham

SUMMARY:
A Randomized, Multi-Center, Pivotal Efficacy and Safety Study Evaluating the RESET System for Glycemic Improvement in Patients with Inadequately Controlled Type 2 Diabetes and Obesity, the STEP-1 Study.

A multi-center, double-blinded, randomized, sham-controlled trial to evaluate the safety and effectiveness of the RESET System plus moderate intensity lifestyle and dietary counseling compliant with 2024 ADA Standard of Care as compared to a sham control receiving moderate intensity lifestyle and dietary counseling. Both the treatment and sham group will practice medical management compliant with STEP-1 Study Guidelines. Patients will be randomized 3 (RESET):1 (Sham).

DETAILED DESCRIPTION:
The objective of this study is to evaluate the safety and effectiveness of the RESET System when used with moderate intensity lifestyle and dietary counseling and medical management, in patients with baseline HbA1c ≥ 7.5% and ≤10%, and BMI ≥ 30 kg/m2 and ≤ 50kg/m2, whose diabetes medications consist of at least dual therapy for 3 months, yet have not achieved adequate HbA1c control (<7%).

Specific objectives of this study are:

1. To determine if the RESET System significantly improves glycemic control
2. To determine that the RESET System can be safely used to improve glycemic control

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥22 years and ≤ 65 years
2. Have understood and signed the approved informed consent form
3. Diagnosis of type 2 diabetes
4. HbA1c ≥ 7.5% and ≤10%
5. BMI ≥30kg/m2 and ≤ 50kg/m2
6. Willing and able to comply with study requirements
7. Documented negative pregnancy test in women of childbearing potential
8. Women of childbearing potential not intending to become pregnant (continue to be on an approved form of birth control) for the duration of their trial participation, including post explant period. Women of child-bearing age without known sterilization will be placed on 1 form of birth-control to prevent unwanted pregnancies
9. At least one year of medical records available, including detailed medical therapy and dosing information
10. Failed to achieve adequate HbA1c reduction (<7.5%) after dual therapy for at least 3-month stable dosage of diabetes medication(s), including insulin, metformin, SGLT-2 inhibitor, GLP-1 RA, Dual GLP-1/GIPR agonist or, other medications including meglitinides, sulfonylureas, thiazolidinediones, or DPP-4s.

Exclusion Criteria:

1. Previous treatment with the RESET System
2. Previous GI surgery that could preclude the ability to place the RESET Liner or affect the function of the RESET Liner, or abnormal GI anatomical finding that could preclude the ability to place the RESET Liner or affect the function of the RESET Liner
3. Hypoglycemia and/or DKA/HHNK in the last 6 months requiring 3rd party assistance
4. Known history of liver disease (e.g., viral or autoimmune etiology, METAVIR grade 2 or higher fibrosis/cirrhosis from a biopsy within the past 6 months, but not including incidental fatty liver)
5. eGFR of less than 45 ml/min/1.73 m2
6. Prior history of an abscess requiring hospitalization, intravenous antibiotics or drainage
7. Previous treatment for severe liver disease and/or biliary tract disease, including but not limited to, surgery, bile duct dilatation, and stent placement
8. Diagnosis of type 1 diabetes mellitus or having any history of ketoacidosis
9. Fasting C-peptide < 1.0 ng/mL
10. Triglyceride level > 600 mg/dL
11. Vitamin D deficiency (<20ng/ml)
12. Uncorrectable bleeding diathesis, platelet dysfunction, thrombocytopenia with platelet count less than 100,000/microliter, or known coagulopathy
13. Height < 5 feet (152.4 cm)
14. Current alcohol addiction, current drug addiction or usage, of drugs such as, narcotics, opiates, or benzodiazepines and other addictive tranquilizers
15. History of pancreatitis, including gallstone related pancreatitis (subsequent to which patient has cholecystectomy)
16. Diagnosis of osteopenia or osteoporosis or currently taking denosumab, romosozumab-aqqg, bisphosphonates or teriparatide
17. Diagnosis of autoimmune connective tissue disorder (e.g. lupus erythematosus, scleroderma)
18. Active or recent (less than 12 months) gastroesophageal reflux disease (GERD) unless treated with H2RAs not PPI.
19. Uncontrolled thyroid disease, including a history of thyroid cancer, hyperthyroidism, or taking thyroid hormone for any reason other than primary hypothyroidism (TSH level must be between 0.4-4)
20. Currently taking prescription antithrombotic therapy (e.g. anticoagulant or antiplatelet agent) within 10 days prior to randomization and/or there is a need or expected need to use during the trial 9 months post implant procedure
21. Currently taking the following medications (within 30 days prior to randomization) and/or there is a need or expected need to use these medications during the trial 12 months post index procedure:

    Restricted Medications/Supplements Systemic corticosteroids Proton Pump Inhibitor (PPI) Drugs known to affect GI motility (e.g.metoclopramide) Prescription or over-the-counter weight loss medication(s) Non-Steroidal Anti-Inflammatory Drugs (NSAIDs), aspirin, ibuprofen, and other anti-inflammatory medication for study duration Medications known to cause significant weight gain or weight loss (e.g. chemotherapeutics)

    Supplements that are known or suspected to increase bleeding risk including but not limited to:

    Gingko biloba Ginseng Vitamins C & E Turmeric St. John's wort Evening primrose oil Feverfew Green Tea Extract
22. Active H. pylori
23. History of Crohn's disease, atresias or untreated stenoses
24. Abnormal pathologies or conditions of the gastrointestinal tract, including ulcers or upper gastrointestinal bleeding conditions within 3 months of randomization
25. Patients may be disqualified for study inclusion for any condition determined by the PI that places the patient at undue risk
26. Poor dentition not allowing complete chewing of food
27. Enrolled in another investigational study within 3 months of screening for this study (enrollment in observational studies is permitted)
28. Residing in a location without ready access to study site medical resources
29. Documented weight loss of 5% total body weight (TBW) anytime during the 3 months preceding randomization
30. Positive Fecal Immunochemical Test (FIT) at time of screening
31. History or observation of psychological disorder or behavior which could preclude compliance to the treatment and follow up plan
32. No access to an active telephone and internet service for provision of Follow Up Schedule calls and electronic diary
33. Having donated blood or received a blood transfusion in the 90 days prior to baseline labs. Patients should agree not to donate blood during the study
34. Any condition that increases red cell turnover, such as thalassemia
35. Existence of (>5 cm string test) Pseudomonas aeruginosa, Stenotrophomonas maltophilia and/or Klebsiella pneumoniae serotype K1 and K2
36. A known sensitivity to nickel or titanium
37. Do not meet the screening criteria for MRI (i.e., MRI unsafe, or MRI conditional but not appropriate for the region of interest)
38. Patients with history or suspicion of coronary artery disease

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2019-09-09 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | 9 Months
  Change in HbA1c value from baseline to 9 months.

SECONDARY OUTCOMES:
HbA1c value | 9 and 21 months
  Proportion of patients who achieve an HbA1c value of < 7 %
Weight Loss | 9 and 21 months
  Proportion of patients who achieve percent total body weight loss ≥ 5% from baseline
Insulin use | 9 and 21 months
  Proportion of patients reducing insulin dosage
LDL cholesterol | 9 and 21 months
  Chnage in LDL cholesterol
Triglycerides | 9 and 21 months
  Change in triglycerides
Blood pressure | 9 and 21 months
  Change in systolic blood pressure values
Fasting blood glucose level | 9 and 21 months
  Change in fasting blood glucose values
Vitamin D | 9 and 21 months
  Change in vitamin D levels
Vitamin D Supplementation | 9 and 21 months
  Average vitamin D levels required to maintain normal vitamin D levels
Refractory to Vitamin D Supplementation | 9 and 21 months
  Proportion of patients refractory to vitamin D supplementation
Serum Creatinine | 9 and 21 months
  Change in serum creatinine levels
eGFR | 9 and 21 months
  Change in eGFR levels
Change in Nonalcoholic Fatty Liver Disease (NAFLD) | 9 and 21 months
  Change in NAFLD, change in % liver fat using MRI (proton density fat fraction)
Change in Nonalcoholic Steatohepatitis (NASH) | 9 and 21 months
  NASH- liver fibrosis % compared to baseline using using MRE measured in kPa
DTSQ Questionnaire | 9 and 21 months
  Change from baseline in treatment satisfaction using Diabetes Treatment Satisfaction Questionnaire (DTSQ)
IWQOL Questionnaire | 9 and 21 months
  Impact of weight on quality of life (IWQOL)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher C Thompson, MD, Principal Investigator — Brigham and Women's Hospital
Locations (7):
- United States (7):
  - MedStar Health Research Institute, Washington D.C., District of Columbia
  - University of Miami Hospital, Miami, Florida
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Michigan Medicine, Division of Gastroenterology and Hepatology, Ann Arbor, Michigan
  - Weill Cornell Medicine, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holman RR, Paul SK, Bethel MA, Matthews DR, Neil HA. 10-year follow-up of intensive glucose control in type 2 diabetes. N Engl J Med. 2008 Oct 9;359(15):1577-89. doi: 10.1056/NEJMoa0806470. Epub 2008 Sep 10. PMID 18784090
- [Background] Rodbard D. Interpretation of continuous glucose monitoring data: glycemic variability and quality of glycemic control. Diabetes Technol Ther. 2009 Jun;11 Suppl 1:S55-67. doi: 10.1089/dia.2008.0132. PMID 19469679
- [Background] Stratton IM, Adler AI, Neil HA, Matthews DR, Manley SE, Cull CA, Hadden D, Turner RC, Holman RR. Association of glycaemia with macrovascular and microvascular complications of type 2 diabetes (UKPDS 35): prospective observational study. BMJ. 2000 Aug 12;321(7258):405-12. doi: 10.1136/bmj.321.7258.405. PMID 10938048
- [Background] Effect of intensive blood-glucose control with metformin on complications in overweight patients with type 2 diabetes (UKPDS 34). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):854-65. PMID 9742977
- [Background] Ford ES, Li C, Little RR, Mokdad AH. Trends in A1C concentrations among U.S. adults with diagnosed diabetes from 1999 to 2004. Diabetes Care. 2008 Jan;31(1):102-4. doi: 10.2337/dc07-0565. Epub 2007 Oct 12. No abstract available. PMID 17934146
- [Background] Detournay B, Cros S, Charbonnel B, Grimaldi A, Liard F, Cogneau J, Fagnani F, Eschwege E. Managing type 2 diabetes in France: the ECODIA survey. Diabetes Metab. 2000 Nov;26(5):363-9. PMID 11119015
- [Background] Mokdad AH, Ford ES, Bowman BA, Dietz WH, Vinicor F, Bales VS, Marks JS. Prevalence of obesity, diabetes, and obesity-related health risk factors, 2001. JAMA. 2003 Jan 1;289(1):76-9. doi: 10.1001/jama.289.1.76. PMID 12503980
- [Background] Torquati A, Lutfi R, Abumrad N, Richards WO. Is Roux-en-Y gastric bypass surgery the most effective treatment for type 2 diabetes mellitus in morbidly obese patients? J Gastrointest Surg. 2005 Nov;9(8):1112-6; discussion 1117-8. doi: 10.1016/j.gassur.2005.07.016. PMID 16269382
- [Background] Rubino F, Gagner M. Potential of surgery for curing type 2 diabetes mellitus. Ann Surg. 2002 Nov;236(5):554-9. doi: 10.1097/00000658-200211000-00003. PMID 12409659
- [Background] Colditz GA, Willett WC, Rotnitzky A, Manson JE. Weight gain as a risk factor for clinical diabetes mellitus in women. Ann Intern Med. 1995 Apr 1;122(7):481-6. doi: 10.7326/0003-4819-122-7-199504010-00001. PMID 7872581
- [Background] Koh-Banerjee P, Wang Y, Hu FB, Spiegelman D, Willett WC, Rimm EB. Changes in body weight and body fat distribution as risk factors for clinical diabetes in US men. Am J Epidemiol. 2004 Jun 15;159(12):1150-9. doi: 10.1093/aje/kwh167. PMID 15191932
- [Background] Ritz E. Limitations and future treatment options in type 2 diabetes with renal impairment. Diabetes Care. 2011 May;34 Suppl 2(Suppl 2):S330-4. doi: 10.2337/dc11-s242. No abstract available. PMID 21525478
- [Background] Aschner P, Kipnes MS, Lunceford JK, Sanchez M, Mickel C, Williams-Herman DE; Sitagliptin Study 021 Group. Effect of the dipeptidyl peptidase-4 inhibitor sitagliptin as monotherapy on glycemic control in patients with type 2 diabetes. Diabetes Care. 2006 Dec;29(12):2632-7. doi: 10.2337/dc06-0703. PMID 17130196
- [Background] Bennett MC, Badillo R, Sullivan S. Endoscopic Management. Gastroenterol Clin North Am. 2016 Dec;45(4):673-688. doi: 10.1016/j.gtc.2016.07.005. PMID 27837781
- [Background] Brethauer SA, Chang J, Galvao Neto M, Greve JW. Gastrointestinal devices for the treatment of type 2 diabetes. Surg Obes Relat Dis. 2016 Jul;12(6):1256-61. doi: 10.1016/j.soard.2016.02.031. Epub 2016 Mar 2. PMID 27568475
- [Background] Frattini F, Borroni G, Lavazza M, Liu X, Kim HY, Liu R, Anuwong A, Rausei S, Dionigi G. New endoscopic procedures for diabetes mellitus type 2 and obesity treatment. Gland Surg. 2016 Oct;5(5):458-464. doi: 10.21037/gs.2016.10.03. PMID 27867859
- [Background] Laubner K, Riedel N, Fink K, Holl RW, Welp R, Kempe HP, Lautenbach A, Schlensak M, Stengel R, Eberl T, Dederichs F, Schwacha H, Seufert J, Aberle J. Comparative efficacy and safety of the duodenal-jejunal bypass liner in obese patients with type 2 diabetes mellitus: A case control study. Diabetes Obes Metab. 2018 Aug;20(8):1868-1877. doi: 10.1111/dom.13300. Epub 2018 Apr 23. PMID 29569313
- See also: Statistics on ASMBS 2016 — http://www.asmbs.org/resources/estimate-of-bariatric-surgery-numbers
- See also: Merck & Co. I. Prescribing information: Januvia (sitagliptin) tablets. 2011:1-23. — http://www.merckconnect.com/januvia/dosing-administration/